CLINICAL TRIAL: NCT04165915
Title: Seniors'Health Paths " PAERPA ", a Support Being Made Available to General Practionners for Assistance in the Management of Elderly Persons at Risk of Losing Their Independence. Review of the Implementation of the Arrangement on the Est-héraultais Territory.
Brief Title: Seniors'Health Paths " PAERPA ",
Acronym: PAERPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0513
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Loss of Autonomy
Keywords: Aged of 60 years and more; living in the Est-Héraultais territory; seniors'health paths; PAERPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
•Background: PAERPA experimentation implemented in the East-Herault region since September 2017 aims to identify fragility and prevent the risk of loss of autonomy in elderly persons older than 60 years by facilitating coordination between Professionals taking care of the patient with the personalized health plan " PPS". The main objective of this study was to evaluate the implementation of this device through the achievement or not of the objectives set by the PPS.

•Methods: Descriptive cohort study with retrospective inclusion and prospective follow-up from the East Herault CTA database. All patients over 60 years old living at home and having a PPS written between September 2017 and April 2018 were included. PPS monitoring for 1 year. Description of this population then analysis of PPS.

•Discussion: Our study aims to evaluate the implementation of the device to identify ways to improve the device for the management of subjects at risk of loss of autonomy.

ELIGIBILITY:
Inclusion Criteria:

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Aged of 60 years and more
* individual health care plan was prepared
* living in the Est-Héraultais territory

Exclusion Criteria:

* Hospitalized patients
* Patients who declined to have an individual heath care planPsychosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient aged 60 and over with an individual health care plan living in the territory of East Heraultais
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Estimating goals set by the PPS (personalized health plan) | 6 and 12 month follow-up
  achievement of objectives established in the individual health care plan after 6 and 12 month follow-up

SECONDARY OUTCOMES:
correlation between unwillingness and cognitive disorder | 1 day
  correlation between unwillingness and cognitive disorder
Correlation between unwillingness and numbers of established goals | 1 day
  Correlation between unwillingness and numbers of established goals
Correlation between unwillingness and locomotors goals | 1 day
  Correlation between unwillingness and locomotors goals

CONTACTS AND LOCATIONS:
Overall Officials: Chokri Boubakri, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC